CLINICAL TRIAL: NCT02133040
Title: Identification and Regulation of Brown Adipose Tissue (BAT) in Humans. Implications for Energy Expenditure in Humans and in the Treatment of Obesity and Related Metabolic Diseases
Brief Title: Effects of Hyperthyroidism on Amount and Activity of Brown Adipose Tissue
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Peter Breining, MD, Aarhus University Hospital
Other Study IDs: M-2013-236-13
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Hyperthyroidism
Keywords: Brown Adipose Tissue
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and fat tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- T3 > 4 nmol/l: Acute hyperthyroidism with a T3 > 4 nmol/l

SUMMARY:
The investigators wish to evaluate the effect of thyroid hormones on brown adipose tissue in humans in an observational study on patients with thyrotoxicosis. In the investigators evaluation the investigators will use FDG-PET/CT, indirect calorimetry and fat biopsies in the acute phase of the disease and in the euthyroid phase after treatment.

It is the investigators hypothesis that high levels of circulating T3 might affect amount and function of brown adipose tissue.

DETAILED DESCRIPTION:
10 patients with thyreotoxicosis (T3 > 3 nmol/L and suppressed TSH) will be investigated at diagnosis and after 3-6 months of euthyroidism induced by antithyroid treatment. The patients will all be over the age of 50 due to the radiation given by the scans (requested by the local Ethical Committee). All will be scanned for active BAT by the integrated FDG PET-CT before and after treatment.BAT is activated by means of crushed ice placed under the feet in individualized intervals during the scan procedure. Indirect calorimetry is done to determine the basal metabolic rate and subcutaneous fat biopsy to examine the effect on subcutaneous white fat and the possible "browning" effect.

ELIGIBILITY:
Inclusion Criteria:

* men and women with hyperthyroidism (T3 > 3 nmol/l)
* > 50 years old
* women must be postmenopausal

Exclusion Criteria:

* thyrotoxic crises
* severe concurrent sickness that will make it unsafe to postpone treatment, this includes severe kidney disease (creatinin over 160)- and heart disease (NYHA group 3 and 4).
* diabetes
* former and current treatment with interleukin-2
* Patients who are already treated with β-blockers
* severe claustrophobia
* BMI > 30 kg/m2

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with hyperthyroidism, reffered to our hospital from their primary caretakers will be investigated before and after 3 to 5 months in a proven euthyroid state.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2020-05-10 (Estimated)

PRIMARY OUTCOMES:
FDG-PET/CT-scanning | 6 months
  Changes in Brown adipose tissue FDG uptake

SECONDARY OUTCOMES:
Indirect Calorimetry | 6 months
  Changes in basal energy expenditure

OTHER OUTCOMES:
Changes in adrenergic receptor status and UCP1, PGC1alpha, PRDM16 and Dio2 levels in subcutaneous fat depots | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Richelsen, Professor, Study Director — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark